CLINICAL TRIAL: NCT01430299
Title: Efficacy and Safety of Integra Accell Evo3 Demineralized Bone Matrix Instrumented Posterolateral Lumbar Spine Fusion
Brief Title: Efficacy and Safety of Accell Evo3 Demineralized Bone Matrix (DBM) in Instrumented Posterolateral Lumbar Spine Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SeaSpine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACC3-US-2010-1
Record Dates: First submitted 2011-08-30; First posted 2011-09-08 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Stenosis; Spondylosis; Degenerative Changes
MeSH Terms: conditions — Constriction, Pathologic; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Demineralized Bone Matrix (Other): a prospective cohort of patients undergoing posterolateral lumbar fusion with Evo3 in the posterolateral space
  Interventions: Device: Demineralized Bone Matrix
- rh-BMP2 (Other): A retrospective cohort of patients who were age- and sex- matched to the prospective cohort who underwent posterolateral lumbar fusion with use of rh-BMP2
  Interventions: Device: rh-BMP2

INTERVENTIONS:
Device: Demineralized Bone Matrix — Accell Evo3 in posteriolateral fusion (prospective cohort)
  Other Names: Accell Evo3
  Arms: Demineralized Bone Matrix
Device: rh-BMP2 — rh-BMP2 in posterolateral fusion (retrospective cohort)
  Other Names: Infuse
  Arms: rh-BMP2

SUMMARY:
The objective of this study is to prospectively evaluate the performance of Integra Accell Evo3 Demineralized Bone Matrix as an adjunct for posterolateral spine fusion with a retrospective comparison to a historical patient cohort.

DETAILED DESCRIPTION:
The objective of this study is to prospectively evaluate the performance of Integra Accell Evo3 Demineralized Bone Matrix as an adjunct for posterolateral spine fusion with a retrospective comparison to a historical patient cohort. The historical patient cohort has not been previously published and therefore, no reference to this group can be provided.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older at the time of surgery
* Require spinal fusion using posterior Transforaminal Lumbar Interbody Fusion (TLIF), Posterolateral Fusion (PLF) or Posterior Lumber Interbody Fusion (PLIF) in 1 to 3 levels between L3-S1
* Follow-up radiographic imaging post surgery

Exclusion Criteria:

* Long term users of medications known to inhibit fusion,bone metabolism or epidural steroid injections
* Immunosuppressive agents, Disease Modifying Anti-rheumatic drugs (DMARDs) or any similar immunomodulating drugs, Growth Factors or Insulin
* Treated with radiotherapy since their surgery
* Medical conditions known to impact bone metabolism, such as Paget's disease, osteoporosis
* Pregnant or lactating women or women wishing to become pregnant
* Prisoner
* Participating in an investigational drug or another device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-06; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Klineberg, M.D., Principal Investigator — University of CA - Davis
Locations (1):
- University of CA-Davis, Dept. of Orthopaedics, Adult & Pediatric Spine Surgery, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- OsteoSurg 300: Prospective study arm: All patients underwent fusion with pedicle screw instrumentation, decortication of dorsal bony elements, and placement of local autograft bone, allograft cancellous chips, and biologic augmentation with OsteoSurge 300 in the posterolateral space.
- rhBMP-2: Retrospective study arm: All patients underwent fusion with pedicle screw instrumentation, decortication of dorsal bony elements, and placement of local autograft bone, allograft cancellous chips, and biologic augmentation with rhBMP-2 in the posterolateral space.
Period: Overall Study
Arm/Group | OsteoSurg 300 | rhBMP-2
Started | 20 | 23
Completed | 16 | 21
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OsteoSurg 300 | rhBMP-2 | Total
Number analyzed (Participants) | 16 | 21 | 37
Age, Customized [Count of Participants; unit: Participants]
  participants over 18 years of age | 16 | 21 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 7 | 13 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 21 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Radiographic Assessments That Indicate Posterolateral Fusion at 12 Months Post Surgery
Description: Posterolateral fusion by radiographic assessment 12 months post surgery
Time Frame: 12 months
Population: One to 3 spinal levels between L3 and S1 were treated per patient. Fusion was assessed twice per treated level. There were 23 OsteoSurge 300 levels and 37 rhBMP-2 levels but 46 OsteoSurge assessments and 74 rhBMP-2 assessments.
Measure: Count of Units; unit: radiographic assessments
Units Other Than Participants: radiographic assessments
Arm/Group | OsteoSurg 300 | rhBMP-2
Number analyzed (Participants) | 16 | 21
Number analyzed (radiographic assessments) | 46 | 74
radiographic assessments | 43 | 74

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | OsteoSurg 300 | rhBMP-2
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/21
Serious Adverse Events (participants affected / at risk) | 5/16 | 3/21
Other Adverse Events (participants affected / at risk) | 9/16 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsteoSurg 300 (N=16) | rhBMP-2 (N=21)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Loss of sensory and/or motor function (Nervous system disorders) | 1 (1) | 0 (0) — decreased sensation in the right lower extremity compared to the left
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Neurologic deficit (Nervous system disorders) | 1 (1) | 0 (0)
Unresolved pain (Nervous system disorders) | 1 (1) | 0 (0) — Patient presents with worsening back pain and new onset radicular symptoms into her right thigh. Also complains of fecal incontinence
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory issues (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient reported 2 days of vomiting and pain radiating from her abdomen to her back. She was diagnosed with symptomatic small bowel volvulus
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsteoSurg 300 (N=16) | rhBMP-2 (N=21)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Fractured Toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dural Tear (Nervous system disorders) | 3 (3) | 4 (4)
Gait disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Loss of sensory and/or motor function (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Numbness/Tingling (Nervous system disorders) | 0 (0) | 1 (1)
Unresolved Pain (Nervous system disorders) | 8 (11) | 9 (14)
Swelling (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombosis (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days